CLINICAL TRIAL: NCT05176249
Title: Lurie Children's Eosinophilic Esophagitis Patient Database
Brief Title: Prospective Database for Eosinophilic Esophagitis (EoE) of Pediatric Population
Acronym: EoE
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Attending Physician, Gastroenterology, Hepatology & Nutrition, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2011-14486
Record Dates: First submitted 2021-10-06; First posted 2022-01-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — 1. Intestinal Biopsies Store in RNAlater or AllProtect
  2. Plasma or Serum from blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophilic Esophagitis (EoE) is a chronic, immune-mediated allergic inflammatory disorder that is being diagnosed with increased frequency. Compelling evidence suggests the etiopathogenesis is allergic and the immune response is triggered by food antigens in most children afflicted with this condition. The literature characterization of EoE is descriptive and retrospective thus far. Our aim in collecting and analyzing data prospectively of all EoE patients seen at Ann & Robert H. Lurie Children's Hospital (Lurie Children's) is to better understand the etiology, pathogenesis and clinical presentation of EoE in patients to better delineate its association with other atopic conditions including reactive airway disease, seasonal allergies and atopic dermatitis. This will allow us to better evaluate the effectiveness of therapeutic strategies used to treat patients with EoE. In addition to collecting data prospectively, the investigators will also review the charts of EoE patients and those suspected of having EoE seen at Lurie Children's. This will allow us to also gather information on control patients, not diagnosed with EoE, who may not be followed in EoE clinic.

DETAILED DESCRIPTION:
Eosinophilic esophagitis has recently emerged as a distinct clinical entity in children and adults. The diagnosis is based on the presence of at least fifteen eosinophils per high power field (hpf) in the esophageal biopsy in children pre-treated with at least eight weeks of adequate acid suppression therapy. The clinical spectrum of EoE varies by age and ranges from failure to thrive and food aversion in toddlers to GERD-like symptoms in school age children to solid food dysphagia and food impaction in adolescents. Although the elemental diet has proven to be more effective than other less restrictive elimination diets in treating EoE, the latter has practical advantages over elemental therapy. In contrast to diet-mediated treatments, topical and systemic corticosteroids are also used to manage EoE symptoms and studies are underway to establish the safety and efficacy of anti-interleukin-5 monoclonal antibodies. The natural history of EoE is not known and prospective studies are needed to understand the etiopathogenesis, distinguish it from other atopic conditions, determine optimal treatment therapies, and to validate noninvasive surrogate tests to monitor histological remission of this enigmatic disorder.

Health outcomes in children and adolescents related to EoE primarily focus on symptoms and histology. This does not take into consideration the health related quality of life (HRQOL), which may be conceptualized to include physical health, mental health, social functioning, role functioning, and general health perceptions. HRQOL has been shown to affect patient satisfaction with and adherence to treatment, and therefore long term outcomes.

The PedsQLTM 4.0 is a, self-administered, non-preference based generic instrument. It consists of a 23-item core measure of global health-related quality of life (HRQOL). The tool includes scales of physical, emotional, social and school function and is validated for children age 2-18 years. Multiple studies have demonstrated the reliability, validity and responsiveness of this instrument in healthy children and in children with chronic diseases. Even more recently developed is the PedsQLTM Eosinophilic Esophagitis Module, a disease-specific tool that has demonstrated excellent feasibility, reliability and validity in EoE patients.

Additionally the investigators are using the Pediatric Eosinophilic Esophagitis Symptom Severity Module, Version 2.0® in measuring patient-relevant outcomes. The 20 question survey was created in an effort to identify and uniquely measure relevant outcomes that patients with EoE and their families identified as important. Within the 20 questions, patient and family input is established from four major domains: dysphagia, gastrointestinal reflux disease (GERD), nausea/vomiting, and pain. A recent study found that the administration of this survey will yield results in the specific domains correlated to specific patient-reported symptoms.

ELIGIBILITY:
Inclusion Criteria:

-Patients with an established diagnosis of EoE, based on endoscopy with biopsies with ≥15 eosinophils per hpf in esophageal biopsies after symptoms of esophageal dysfunction persist despite at least 6-8 weeks of appropriate acid suppression therapy.

OR

-Patients who are suspected of having EoE (presenting with symptoms of esophageal dysfunction non-responsive to appropriate proton pump inhibitor therapy for 6-8 weeks).

• Note: Patients suspected of having EoE but not diagnosed with EoE by endoscopy with biopsies will serve as control patients

Exclusion Criteria:

* Patients who do not consent to participate

Ages: 1 Month to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Study population is determined through general GI and EOE specific clinics. Patients who are undergoing pre-diagnostic endoscopies to change of treatments are enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Perform a prospective analysis of all the EoE patients as well as patients suspected of having EoE | estimated every 6-12 months; at time of all standard of care endoscopies
  to compare the efficacy of the different treatment modalities used in these patients to study the natural history of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Dellon ES, Jensen ET, Martin CF, Shaheen NJ, Kappelman MD. Prevalence of eosinophilic esophagitis in the United States. Clin Gastroenterol Hepatol. 2014 Apr;12(4):589-96.e1. doi: 10.1016/j.cgh.2013.09.008. Epub 2013 Sep 11. PMID 24035773
- [Background] Soon IS, Butzner JD, Kaplan GG, deBruyn JC. Incidence and prevalence of eosinophilic esophagitis in children. J Pediatr Gastroenterol Nutr. 2013 Jul;57(1):72-80. doi: 10.1097/MPG.0b013e318291fee2. PMID 23539047
- [Background] Ingle SB, Patle YG, Murdeshwar HG, Pujari GP. A case of early eosinophilic gastroenteritis with dramatic response to steroids. J Crohns Colitis. 2011 Feb;5(1):71-2. doi: 10.1016/j.crohns.2010.10.002. Epub 2010 Dec 18. No abstract available. PMID 21272810
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Franciosi JP, Hommel KA, Bendo CB, King EC, Collins MH, Eby MD, Marsolo K, Abonia JP, von Tiehl KF, Putnam PE, Greenler AJ, Greenberg AB, Bryson RA, Davis CM, Olive AP, Gupta SK, Erwin EA, Klinnert MD, Spergel JM, Denham JM, Furuta GT, Rothenberg ME, Varni JW. PedsQL eosinophilic esophagitis module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2013 Jul;57(1):57-66. doi: 10.1097/MPG.0b013e31828f1fd2. PMID 23478422
- [Background] Franciosi JP, Hommel KA, DeBrosse CW, Greenberg AB, Greenler AJ, Abonia JP, Rothenberg ME, Varni JW. Development of a validated patient-reported symptom metric for pediatric eosinophilic esophagitis: qualitative methods. BMC Gastroenterol. 2011 Nov 18;11:126. doi: 10.1186/1471-230X-11-126. PMID 22099448
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Varni JW, Seid M, Smith Knight T, Burwinkle T, Brown J, Szer IS. The PedsQL in pediatric rheumatology: reliability, validity, and responsiveness of the Pediatric Quality of Life Inventory Generic Core Scales and Rheumatology Module. Arthritis Rheum. 2002 Mar;46(3):714-25. doi: 10.1002/art.10095. PMID 11920407
- [Background] Martin LJ, Franciosi JP, Collins MH, Abonia JP, Lee JJ, Hommel KA, Varni JW, Grotjan JT, Eby M, He H, Marsolo K, Putnam PE, Garza JM, Kaul A, Wen T, Rothenberg ME. Pediatric Eosinophilic Esophagitis Symptom Scores (PEESS v2.0) identify histologic and molecular correlates of the key clinical features of disease. J Allergy Clin Immunol. 2015 Jun;135(6):1519-28.e8. doi: 10.1016/j.jaci.2015.03.004. PMID 26051952